CLINICAL TRIAL: NCT03589638
Title: Effects of C-MAC Videolaryngoscope, McGRATH Videolaryngoscope and Macintosh Direct Laryngoscope on Intraocular Pressure and Hemodynamics; a Randomized, Double-blind Clinical Trial
Brief Title: Effects of C-MAC Videolaryngoscope, McGRATH Videolaryngoscope and Macintosh Direct Laryngoscope on Intraocular Pressure and Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, Department of anesthesia, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asozkan 6
Record Dates: First submitted 2018-06-18; First posted 2018-07-18 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Anesthesiology Devices Associated With Adverse Incidents; Intraocular Pressure
Keywords: tracheal intubation; videolaryngoscopy; hemodynamics; intraocular pressure

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, double blind Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- direct laryngoscope (Active Comparator): Endotracheal intubation was applied by anesthesiologist with direct laryngoscope.
  Interventions: Device: Direct laryngoscope; Device: C-MAC videolaryngoscope; Device: McGrath videolaryngoscope
- C-MAC videolaryngoscope (Active Comparator): Endotracheal intubation was applied by anesthesiologist with C-MAC videolaryngoscope.
  Interventions: Device: Direct laryngoscope; Device: C-MAC videolaryngoscope; Device: McGrath videolaryngoscope
- McGrath videolaryngoscope (Active Comparator): Endotracheal intubation was applied by anesthesiologist with McGrath videolaryngoscope.
  Interventions: Device: Direct laryngoscope; Device: C-MAC videolaryngoscope; Device: McGrath videolaryngoscope

INTERVENTIONS:
Device: Direct laryngoscope — Endotracheal intubation was applied by anesthesiologist wtih direct laryngoscope. SAP (systolic arterial pressure), DAP (diastolic arterial artery pressure), MAP (mean arterial pressure) were measured before and 5 minutes after intubation, , Heart rate (HR), SPO2 (oxygen saturation by pulse oximetry), PI (perfusion index), and intraocular pressure values measured by the eye clinician using the device.
Device: C-MAC videolaryngoscope — Endotracheal intubation was applied by anesthesiologist wtih direct laryngoscope. SAP (systolic arterial pressure), DAP (diastolic arterial artery pressure), MAP (mean arterial pressure) were measured before and 5 minutes after intubation, , Heart rate (HR), SPO2 (oxygen saturation by pulse oximetry), PI (perfusion index), and intraocular pressure values measured by the eye clinician using the device.
Device: McGrath videolaryngoscope — Endotracheal intubation was applied by anesthesiologist wtih direct laryngoscope. SAP (systolic arterial pressure), DAP (diastolic arterial artery pressure), MAP (mean arterial pressure) were measured before and 5 minutes after intubation, , Heart rate (HR), SPO2 (oxygen saturation by pulse oximetry), PI (perfusion index), and intraocular pressure values measured by the eye clinician using the device.

SUMMARY:
In this study, participants aimed to compare the effects of direct laryngoscopic endotracheal intubation and videolaryngoscopic intubation with C-MAC videolaryngoscope and McGrath videolaryngoscope on intraocular pressure and hemodynamics.

DETAILED DESCRIPTION:
The maintenance of airway opened is one of the main responsibility of the anesthetist. Intubation procedure during anesthesia application benefits such as airway opening, airway and breathing control, aspiration hazard, respiratory effort and dead space reduction, surgical comfort and airway control during resuscitation. Laryngoscopy and tracheal intubation increases in heart rate, blood pressure and the intraocular pressure. The sympathetic-adrenal activity caused by the stimulation of the laryngeal and tracheal tissues is responsible for these negative effects. Endotracheal intubation with videolaryngoscopy is an alternative method used in airway management. Laryngoscopy and tracheal intubation under general anesthesia and laryngeal mask and airway control techniques cause different hemodynamic and catecholamine levels.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Score 1-2
* Mallampati 1 ve 2

Exclusion Criteria:

* Glaucoma,
* Diabetes mellitus
* Cardiovascular and pulmonary disease
* American Society of Anesthesiologist Score III-IV
* Bdoy mass index greater than 35
* Difficult intubation history
* Obstetric surgery
* Propofol, fentanyl, rocuronium contraindication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65 years
Enrollment: 3 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.

SECONDARY OUTCOMES:
mean arterial pressure | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.
systolic arterial pressure | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.
diastolic arterial pressure | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.
heart rate | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.
peripheral oxygen saturation | From beginning of Anesthesia to 10th minute of surgery
  The relevant values will be measured in the determined time.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Selim Ozkan, MD, Principal Investigator — İnönü Üniversitesi Tıp Fakültesi
Locations (1):
- Inonu University Medical Faculty, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No